CLINICAL TRIAL: NCT02881411
Title: Self Soft Tissue Therapy for Fibromyalgia Syndrome; Randomised Controlled Feasibility Study
Brief Title: Self Soft Tissue Therapy for Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Royal United Hospital Bath NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JMA/It
Record Dates: First submitted 2016-08-10; First posted 2016-08-29 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Fibromyalgia Syndrome
Keywords: self-soft tissue therapy; trigger points; feasibility study
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-soft tissue therapy (Active Comparator): Intervention group: Fibromyalgia coping skills programme plus self-soft tissue therapy (SSTT) SSTT consists of MTrP therapy on TrP sites in either the lower leg/foot or forearm/hand. MTrP therapy will be administered by the researcher for only two sessions which will include training to teach the participant how to do SSTT on themselves. All participants in the intervention group will also receive an advice booklet for SSTT.
  Interventions: Other: Self-soft tissue therapy
- Fibromyalgia coping skills programme (Active Comparator): Control group:Fibromyalgia coping skills programme only. The FCSP is a non-pharmacological, multidisciplinary exercise and education group programme. Its main aims are to provide condition-specific, patient centred, self-management education and advice, in line with national drivers for long-term conditions and international FMS clinical guidelines.
  Interventions: Other: Fibromyalgia coping skills programme

INTERVENTIONS:
Other: Self-soft tissue therapy — Manual therapy for the muscles in the upper or lower limbs.
  Arms: Self-soft tissue therapy
Other: Fibromyalgia coping skills programme — Exercise, education programme
  Arms: Fibromyalgia coping skills programme

SUMMARY:
The main aims of this preliminary research are to determine if combined self-soft tissue therapy (SSTT) alongside an established 6 week FMS Coping Skills Programme (FCSP) is a feasible and acceptable treatment approach for FMS. All participants on the six week FCSP will be randomly allocated to a control (FMS Coping Skills Programme) or intervention group (FMS Coping Skills Programme plus SSTT). All participants will be assessed for outcome measurements at the start of the feasibility study, at six weeks and three months after completion.

This feasibility study hypothesis is that the SST approach will be acceptable to FMS patients and that the combined 6 week FCSP (hands off) and SSTT (hands on) will be beneficial. This feasibility study will inform a larger randomized controlled trial (RCT) on this combined treatment approach to FMS.

DETAILED DESCRIPTION:
AIMS & OBJECTIVES

The main aims of this preliminary research are:

1. To determine the feasibility of conducting a future larger study in terms of recruitment, randomisation, estimates of effect size, study protocol and procedure, intervention and outcome acceptability.
2. To determine if combining SSTT (MTrP therapy) as an adjunct to the presently only provided usual care of hands off (rehabilitation and self-management programme) is feasible and acceptable to participants in this combined treatment approach to FMS.

METHOD

The multidisciplinary team includes researchers and health professionals who are actively involved in musculoskeletal therapy and research. This current randomised controlled feasibility study is supported by internal funding from the Faculty of Health & Applied Sciences, University of the West of England (UWE), Bristol. Ethics approval from NHS ethics/IRAS has been obtained.

Participant be identification and recruitment Participants will be identified and recruited from those FMS patients enrolled on the 6 week FCSP in the Royal National Hospital for Rheumatic Diseases (RNHRD) out-patients department. All enrolled patients on the FCSP, will be emailed and sent out an invitation letter and information sheet by the RNHRD admin and clinical team requesting participation in the feasibility study.

Prior to primary collection of data, all participants sign an informed consent form. Participants will undergo a screening (for inclusion/exclusion criteria), will provide demographic information and complete a general health screening survey.

Randomisation- All participants will be randomly allocated to either a control or intervention group, by an independent researcher using block randomisation utilising an online randomisation tool. This method involves creating a table using two number sets. The randomiser ensures each group appears an equal number of times whilst simultaneously randomly allocating participants to each group. The randomisation order will be performed by the co-researcher, who will prepare opaque envelopes that can be opened at a relevant point in the process.

Control Group - Participants will undertake the 6 FCSP only. The FCSP is a non-pharmacological, multidisciplinary exercise and education group programme. Its main aims are to provide condition-specific, patient centred, self-management education and advice, in line with national drivers for long-term conditions and international FMS clinical guidelines.

All group participants are screened prior to acceptance onto the FCSP and must have a diagnosis of fibromyalgia using the ACR 1990 or 2010 criteria. Patients with co-morbidities are accepted. Core components of the 6 week FCSP include goal-setting, pacing, hydrotherapy, exercise and dietary advice. There is one face-to-face review session three months after the taught component of the FCSP is completed.

Patient reported outcome measures (PROMS) are collected from participants at three time-points; start of course, end of course and three months post course. These are inputted onto a clinical database, and analysed to measure clinical progress on an individual basis

Intervention Group - Participants in this group will undertake the 6 week FCSP plus SSTT (myofascial trigger point (MTrP) therapy) (initially TrP pressure release performed by the researcher and then also taught a SSTT home programme). The specific form of soft tissue therapy used in this feasibility study is MTrP therapy, as used in a case series on triceps surae dysfunction as described in the protocol below. This protocol is adapted for patients with FMS and will be administered by the researcher for only two sessions which will include training to teach the participant how to do SSTT on themselves. All participants in the control group will receive an advice booklet for SSTT.

Researcher TrP pressure release intervention- Lower leg/foot- The participants will be positioned prone with the knee extended for TrP pressure release on the gastrocnemius and knee flexed for the soleus. While still in prone, TrP pressure release will also be used on the medial plantar aspect of the foot specifically quadratus plantar and abductor halluces. TrP pressure release, employing the barrier release concept will be used. The researcher will slowly apply increasing thumb pressure on the soleus or gastrocnemius MTrPs until the first increase in tissue resistance is felt (barrier). Pressure will initially be perceived as tender or mildly painful, but participants will be instructed to notify the researcher to stop if the procedure is not tolerable. Pressure will be maintained until a release in muscle tension or until the participant feels no tenderness or pain only related to the thumb pressure. On releasing the pressure the researcher will apply a passive stretch to the affected calf muscle, to facilitate maintenance of the gained muscle length. On subsequent visits TrP pressure release will be progressed while rocking or facilitating the ankle into greater dorsiflexion and will be applied to the hamstrings while flexing and extending the knee. Participants will be warned about possible mild post treatment soreness (mild ache) which may last up to 24 hours, but will not interfere with day to day function.

Forearm/Hand- Exactly the same TrP pressure release protocol will be used. All participants will be seated with the forearm resting on a plinth, with researcher and participant facing each other. The thenar and hypothenar muscles, wrist extensor and flexor muscles will receive TrP pressure release and stretching.

Self soft tissue therapy (SSTT)- participants will be advised on self treatment and shown the technique on identified active or latent MTrPs in the lower leg/foot or forearm/hand. Participants will be shown varying techniques including self-massage, use of a tennis ball or foam roller. All participants will be advised to do SSTT at least once a day and advised to stop SSTT if symptoms are increased.

Stretching programme - stretching is advised post SSTT of MTrPs as part of a home exercise programme. A standardised home stretching protocol will be issued and detailed in the advice booklet including demonstration of the stretching techniques and advice on dosage. A full description and demonstration will be given to participants. No specific time will be given for the stretching protocol as the evidence is inconclusive on the duration of static stretch needed to produce benefit.

Data management and analysis- Data will be analysed by the PI and co-researcher in an office at the University of the West of England. Statistical Package for the Social Sciences (SPSS) version 20.0 will be used to analyse the data using descriptive (mean, standard deviation and range of scores at the initial and follow up sessions). The results of the additional FCSP /FMS PROMS and criteria for FMS diagnosis-Widespread Pain Index/Symptom Severity Score plus tenderness in 18 tender point sites will also be analysed for differences between groups. In line with the aims of this feasibility study, no inferential statistics will be employed.

Sampling frame-

As this is feasibility study no sample size or power calculation has been conducted. The aim is to recruit 20 patients, enough to meet the aims of a feasibility study and being sufficient to provide estimates of variability between the control and intervention groups. All potential participants to be screened and accepted if they meet the inclusion/exclusion criteria:

Confidentiality/ Anonymity- Any data produced from the feasibility study will be anonymised; therefore, any identifying details will be replaced numerically. All data will be analysed and downloaded on a password protected computer at the University of the West of England.

Data handling and Record Keeping- The CI and PI will be responsible for data collection, recording and quality. Anonymised collected data from each participant will be analysed and downloaded on a password protected computer at the University of the West of England. Data will be collected and retained in accordance with the Data Protection Act 1998. Back-up copies of electronic data will be made regularly onto a CD. All source documents will be retained for a period of 5 years following the end of the study.

Addressing Consent & Withdrawal- Consent- Consent will be addressed via an informed consent form that will be given to all participants a week before data collection and signed prior to collection of data. A full explanation and opportunity to ask questions prior and during data collection will be afforded to all participants.

Withdrawal- Participants are completely free to abstain or withdraw from the feasibility study at any time during the process of data collection.

Risk & Risk Management- Participants will be invited to participate in the feasibility study. Each participant will have the option to participate or opt out. Participants' futures will not be affected in any way by their decision to take part or not. There will not be any physical, psychological, social legal or economic risks for participants to participate in the feasibility study. There will be no additional risks to the researchers or other people impacted by this study as a consequence of undertaking this proposal that are greater than those encountered in normal day-to-day life.

Access to source data- Direct access to the source data and documents will be permitted for monitoring, audits, Research Ethics Committees and review.

Safety Assessments and Monitoring- The project management committee will consist of the research team (Dr Rob Grieve, Sandi Derham and Julie Russell), who will meet regularly to assess the study. This study will be monitored and audited in accordance with UWE policy.

Other Ethical Considerations- Apart from the already mentioned possible mild discomfort, participants will have to make an effort to attend the sessions and do the SSTT home programme.

ELIGIBILITY:
Inclusion Criteria:

Aged over 18. Able be seated or lie prone for 30 minutes. Diagnosis or presentation of FMS and attending FMS coping skills programme. Complaint of forearm/hand or lower leg/foot pain or tenderness for the past 7 days..

No disorder apart from FMS, that would otherwise explain the pain or tenderness..

Exclusion criteria:

Complex regional pain syndrome. Talipes equino varus, triple arthrodesis. Bony block of the ankle. Lower leg/foot injury. Forearm/hand injury. Diabetes. Peripheral vascular disease. Cancer. Rheumatoid arthritis or neurological impairment. Receiving physiotherapy or MTrP therapy to the upper or lower limb within the previous three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT)-Change is being assessed. | Baseline day 0, conclusion at 6 weeks and three months after conclusion
  Algometry of myofascial trigger points

SECONDARY OUTCOMES:
Verbal Numerical Rating Scale-Verbal description of pain from 0-10-Change is being assessed | Baseline day 0, conclusion at 6 weeks and three months after conclusion
  Participants indicate the intensity of pain by reporting a number that best represents it, between 0 (no pain) and 10 (maximum pain).
Range of Movement (ROM)-Change is being assessed. | Baseline day 0, conclusion at 6 weeks and three months after conclusion
  Goniometric measurements for ankle and wrist
Disabilities of Arm, Shoulder and Hand (DASH)-30-item, self-report questionnaire- Change is being assessed. | Baseline day 0, conclusion at 6 weeks and three months after conclusion
  Is a validated standardised measure of physical function and symptoms in patients with musculoskeletal disorders of the upper limb.
Lower Extremity Functional Scale (LEFS)-self-reported questionnaire (0-80 points)-Change is being assessed | Baseline day 0, conclusion at 6 weeks and three months after conclusion
  Is a validated standardised measure of lower limb function. A change in LEFS scores of 9 points or greater is a true change (CI 90%) and also a clinically meaningful functional change

CONTACTS AND LOCATIONS:
Overall Officials: Rob M Grieve, PhD, Principal Investigator — University of the West of England
Locations (1):
- Royal National Hospital for Rheumatic Diseases (RNHRD), Bath, NE Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data of individual participants will be made available in the results section of a publication. Anonymous data will be presented in the form of descriptive statistics in table or text format.

REFERENCES:
- [Background] Grieve R, Barnett S, Coghill N, Cramp F. Myofascial trigger point therapy for triceps surae dysfunction: a case series. Man Ther. 2013 Dec;18(6):519-25. doi: 10.1016/j.math.2013.04.004. Epub 2013 Jun 5. PMID 23756031
- [Background] Renan-Ordine R, Alburquerque-Sendin F, de Souza DP, Cleland JA, Fernandez-de-Las-Penas C. Effectiveness of myofascial trigger point manual therapy combined with a self-stretching protocol for the management of plantar heel pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2011 Feb;41(2):43-50. doi: 10.2519/jospt.2011.3504. Epub 2011 Jan 31. PMID 21285525
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- See also: Randomization Tool — http://www.randomizer.org/